CLINICAL TRIAL: NCT03352427
Title: A Phase 2 Study of Dasatinib in Combination With Everolimus for Children With Gliomas Harboring PDGFR Alterations
Brief Title: Study of Dasatinib in Combination With Everolimus for Children and Young Adults With Gliomas Harboring Platelet-Derived Growth Factor Receptor (PDGFR) Alterations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.042; HUM00123094 (Other: University of Michigan)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Glioma; High Grade Glioma; Pontine Tumors
MeSH Terms: conditions — Glioma; Brain Stem Neoplasms | interventions — Dasatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib+Everolimus (Experimental): Dasatinib = 60 mg/m2 orally twice daily
  Everolimus = starting dose of 3.0 mg/m2, with titration of dosing after first cycle to keep everolimus trough level of 5-15 ug/ml
  Both agents will be taken daily for 28 day cycles. Cycles will be repeated every 28 days and patients may receive up to 24 cycles.
  Interventions: Drug: Dasatinib; Drug: Everolimus

INTERVENTIONS:
Drug: Dasatinib — 60 mg/m2 orally twice daily
Drug: Everolimus — 3.0 mg/m2, with titration of dosing after first cycle to keep trough level of 5-15 ug/ml

SUMMARY:
This trial will evaluate the activity of dasatinib in combination with everolimus for children with gliomas harboring PDGFR alterations, including newly diagnosed high-grade glioma (HGG) or diffuse intrinsic pontine glioma (DIPG) after radiation (stratum A); and recurrent/progressive glioma (grade II-IV, including DIPG) (stratum B).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of a newly diagnosed high-grade glioma or diffuse intrinsic pontine glioma (DIPG) (Stratum A)
* Histological confirmation (at diagnosis or relapse) of a recurrent or progressive grade II-IV glioma (including DIPG) (Stratum B)
* Participants must have a genomic (DNA and/or RNA) alteration (mutation, fusion, and/or amplification) involving PDGF-A, PDGF-B, PDGFR-A or PDGFR-B, as identified by tumor sequencing.
* Age at enrollment: Greater than 1 year and less than 50 years
* BSA (body surface area): BSA greater than 0.3 m2
* Karnofsky (Measure of performance for cancer patients where 100% represents perfect health) > 50% for patients > 16 years of age and Lansky (Measure of performance for pediatric cancer patients where 100% represents perfect health) > 50% for patients < 16 years of age. Neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 7 days. Patients who are unable to walk because of paralysis, but who are able to sit in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate bone marrow function per protocol
* Adequate liver function per protocol
* Adequate renal and metabolic function per protocol
* Patients with known seizure disorder must have seizures adequately controlled with non- enzyme inducing antiepileptic medications
* No increase in steroid dose within the past 7 days
* Primary brain or spine tumor are eligible, including tumors with metastases, multiple lesions.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy.
* Myelosuppressive chemotherapy: Must not have received within 3 weeks.
* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor, 14 days for long- acting.
* Biologic (anti-neoplastic agent): At least 7 days or 3 half-lives (whichever is longer) since the completion of therapy.
* Radiation therapy:

  * Stratum A: ≥ 2 weeks and </= to 12 weeks must have elapsed from radiation.
  * Stratum B: ≥ 2 weeks must have elapsed from focal radiation.
* > 3 weeks from major surgery. If recent craniotomy, adequate wound healing must be determined by neurosurgical team.
* Autologous Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 4 weeks must have elapsed.
* All patients and/or a legal guardian must sign institutionally approved written informed consent and assent documents.

Exclusion Criteria:

* Patients who are breastfeeding, pregnant or refuse to use an effective form of birth control are excluded.
* Patients with uncontrolled infection are excluded.
* Patients receiving other anti-neoplastic agents are excluded.
* Patients requiring strong CYP3A4 or PGP inhibitors are excluded (per protocol)
* Patients requiring anticoagulation or with uncontrolled bleeding are excluded.
* Patients on steroids for symptom management must be on a stable dose for 7 days prior to start of treatment.
* Patients within 1 year of allogeneic stem cell transplant, patients with active GVHD or requiring immunosuppression are excluded.
* Previous hypersensitivity to rapamycin or rapamycin derivatives

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Koschmann, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miklja Z, Yadav VN, Cartaxo RT, Siada R, Thomas CC, Cummings JR, Mullan B, Stallard S, Paul A, Bruzek AK, Wierzbicki K, Yang T, Garcia T, Wolfe I, Leonard M, Robertson PL, Garton HJ, Wahl DR, Parmar H, Sarkaria JN, Kline C, Mueller S, Nicolaides T, Glasser C, Leary SE, Venneti S, Kumar-Sinha C, Chinnaiyan AM, Mody R, Pai MP, Phoenix TN, Marini BL, Koschmann C. Everolimus improves the efficacy of dasatinib in PDGFRalpha-driven glioma. J Clin Invest. 2020 Oct 1;130(10):5313-5325. doi: 10.1172/JCI133310. PMID 32603316

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dasatinib+Everolimus
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 10 [4 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in Participants With Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG)
Description: Percentage of participants without progression, defined as 25% increase in the size of the tumor or appearance of new lesions.
Time Frame: 8 months
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
percentage of participants | 0

2. Primary Outcome: Progression-free Survival in Participants With Newly Diagnosed High-grade Glioma (HGG)
Description: as for outcome 1
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
percentage of participants | 0

3. Primary Outcome: Overall Response Rate (OR) (Partial Response or Better) in Participants With Refractory or Recurrent Glioma
Description: The overall response assessment will take into account response in both target and non-target lesions, as well as the appearance of new lesions. Partial Response (PR) will be defined as ≥50% decrease in size of tumor in comparison to baseline measurements. Complete Response (CR) will be defined as the disappearance of all abnormal signal. This includes return to normal size of the brain stem for brain stem lesions. Reported as percentage of participants with partial or better response at 56 days.
Time Frame: 56 Days
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
percentage of participants | 0

4. Secondary Outcome: Overall Survival
Description: Percentage of patients alive at one year.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
percentage of participants | 0

5. Secondary Outcome: Overall Survival
Description: Percentage of participants alive at 2 years.
Time Frame: up to 17 months
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib+Everolimus
Number analyzed (Participants) | 3
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days after the last dose of study treatment (total of 17 months; average of 4 months). All cause mortality occurred any time during the study (range from 4 - 17 months).
Arm/Group | Dasatinib+Everolimus
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib+Everolimus (N=3)
headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib+Everolimus (N=3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Eye disorders (Eye disorders) | 1
Dysarthria (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Fatigue (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Ataxia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Edema face (General disorders) | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 — Left ear clogged, Gr 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
tremor (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 1
Flushing (Vascular disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1

LIMITATIONS AND CAVEATS:
Trial enrollment was limited due to requirement for patient insurance coverage for all aspects of treatment. Due to limited sample size, full statistical analysis isn't possible. Descriptive results of this cohort compiled with data available from patients treated locally with a similar treatment plan is available in the following publication: Miklja et al, JCI, 2020 [PMID: 32603316].

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03352427/Prot_SAP_000.pdf